CLINICAL TRIAL: NCT01457677
Title: A Multi Center, Randomized, Double-blind, Placebo Controlled, Parallel-group Study to Investigate the Efficacy and Safety of RO4995819 Versus Placebo, as Adjunctive Therapy in Patients With Major Depressive Disorder Having Inadequate Response to Ongoing Antidepressant Treatment (ARTDeCo)
Brief Title: ARTDeCo Study: A Study of RO4995819 in Patients With Major Depressive Disorder And Inadequate Response to Ongoing Antidepressant Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BP25712
Record Dates: First submitted 2011-10-20; First posted 2011-10-24 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- RO4995819 15 mg (Experimental)
  Interventions: Drug: RO4995819
- RO4995819 30 mg (Experimental)
  Interventions: Drug: RO4995819
- RO4995819 5 mg (Experimental)
  Interventions: Drug: RO4995819

INTERVENTIONS:
Drug: Placebo — matching placebo to RO4995819 oral once daily for 6 weeks
  Arms: Placebo
Drug: RO4995819 — 5 mg oral once daily for 6 weeks
  Arms: RO4995819 5 mg
Drug: RO4995819 — 15 mg oral once daily for 6 weeks
  Arms: RO4995819 15 mg
Drug: RO4995819 — 30 mg oral once daily for 6 weeks
  Arms: RO4995819 30 mg

SUMMARY:
This multi-center, randomized, double-blind, placebo-controlled, parallel-group study will investigate the efficacy and safety of RO4995819 as adjunctive therapy in patients with major depressive disorder having inadequate response to ongoing antidepressant treatment. Patients will be randomized to receive once daily doses of 5 mg, 15 or 30 mg of RO4995819 or matching placebo. The anticipated time on study treatment is 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, 18-65 years of age
* Major depression disorder without psychotic features
* Inadequate response to current, ongoing antidepressant treatment as defined by protocol
* Having at least one but no more than 2 antidepressant treatment trial failures
* Body mass index (BMI) 18.0-35.0 kg/m2 inclusive

Exclusion Criteria:

* Patient currently receives treatment with a combination of 3 or more antidepressants
* Significant ongoing use of high doses of barbiturates, benzodiazepines or other anxiolytic drugs
* Patient previously received RO4995819
* Patient participated in an investigational drug or device trial within 6 months of screening
* History of non-response to, or current use of non-pharmacological treatment including Electroconvulsive Therapy (ECT), Vagus Nerve Stimulation (VNS), or Repetitive Transcranial Magnetic Stimulation (RTMS)
* Past or present psychotic symptoms

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 357 (Actual)
Dates: Start 2011-12; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Mean change in Montgomery Asberg Depression Rating Scale (MADRS) scores | 6 weeks

SECONDARY OUTCOMES:
Safety (incidence of a adverse events) | 6 weeks
Proportion of patients exhibiting remission based on the Montgomery Asberg Depression Rating Scale (MADRS) (score of </=10) | 6 weeks
Proportion of patients exhibiting response based on the Montgomery Asberg Depression Rating Scale (MADRS) (reduction in score of >/= 50% of the baseline score) | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (82):
- United States (40):
  - Phoenix, Arizona
  - Oakland, California
  - Redlands, California
  - San Diego, California
  - Stanford, California
  - Torrance, California
  - Victorville, California
  - Denver, Colorado
  - Coral Springs, Florida
  - Gainsville, Florida
  - Jacksonville, Florida
  - Lauderhill, Florida
  - North Miami, Florida
  - Ocala, Florida
  - Atlanta, Georgia
  - Roswell, Georgia
  - Smyrna, Georgia
  - Chicago, Illinois
  - Prairie Village, Kansas
  - Wichita, Kansas
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Watertown, Massachusetts
  - Flowood, Mississippi
  - O'Fallon, Missouri
  - Albuquerque, New Mexico
  - New York, New York
  - Rochester, New York
  - Durham, North Carolina
  - Beachwood, Ohio
  - Canton, Ohio
  - Cincinnati, Ohio
  - Jenkintown, Pennsylvania
  - Media, Pennsylvania
  - Columbia, South Carolina
  - Arlington, Texas
  - Houston, Texas
  - Salt Lake City, Utah
  - Richmond, Virginia
  - Roanoke, Virginia
- Austria (3):
  - Innsbruck
  - Vienna
  - Wien, Vienna
- Canada (6):
  - Kentville, Nova Scotia
  - Kingston, Ontario
  - Ottowa, Ontario
  - Gatineau, Quebec
  - Sherbrooke, Quebec
  - Verdun, Quebec
- Germany (7):
  - Ellwangen
  - Leipzig
  - Mannheim
  - Nuremberg
  - Oranienburg
  - Ostfildern
  - Schwerin, Mecklenburg-Vorpommern
- Russia (10):
  - Lipetsk
  - Moscow
  - Novosibirsk
  - Saint Petersburg
  - Samara
  - Smolensk
  - Talagi
  - Tomsk
  - Yaroslavl
  - Yekaterinburg
- Slovakia (3):
  - Bratislava
  - Rimavská Sobota
  - Trenčín
- South Africa (5):
  - Bellville, Cape Town
  - Cape Town, Western Cape
  - Cape Town, Western CAPE
  - Centurion, Pretoria
  - Nieu Muckleneuk, Pretoria
- Ukraine (8):
  - Dnipropetrovsk
  - Donetsk
  - Kharkiv
  - Kherson,Vil. Stepanivka
  - Kiev
  - Odesa
  - Simferopol, Crimea
  - Vinnytsia

REFERENCES:
- [Derived] Dean RL, Hurducas C, Hawton K, Spyridi S, Cowen PJ, Hollingsworth S, Marquardt T, Barnes A, Smith R, McShane R, Turner EH, Cipriani A. Ketamine and other glutamate receptor modulators for depression in adults with unipolar major depressive disorder. Cochrane Database Syst Rev. 2021 Sep 12;9(9):CD011612. doi: 10.1002/14651858.CD011612.pub3. PMID 34510411
- [Derived] Umbricht D, Niggli M, Sanwald-Ducray P, Deptula D, Moore R, Grunbauer W, Boak L, Fontoura P. Randomized, Double-Blind, Placebo-Controlled Trial of the mGlu2/3 Negative Allosteric Modulator Decoglurant in Partially Refractory Major Depressive Disorder. J Clin Psychiatry. 2020 Jul 14;81(4):18m12470. doi: 10.4088/JCP.18m12470. PMID 32663909